CLINICAL TRIAL: NCT06266260
Title: Evaluation of Direct Portal Pressure Measurement by Endoscopic Ultrasound in Advanced Chronic Liver Disease and Newly Diagnosed Clinically Significant Portal Hypertension (EVADIPP)
Brief Title: Direct Portal Pressure Measurement Via Endoscopic Ultrasound in Advanced Chronic Liver Disease (EVADIPP)
Acronym: EVADIPP
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Santopaolo Francesco, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5486
Record Dates: First submitted 2023-09-11; First posted 2024-02-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EUS PPG measurement — Direct EUS PPG measurement

SUMMARY:
A minimally invasive procedure to directly assess portal pressure gradient under endoscopic ultrasound guidance (EUS-PPG) has become available and initial data have proved the technique to be safe. Aims of our proposal are: (i) to assess performance of EUS-PPG as compared to HVPG in evaluating hemodynamic response to non selective betablockers (NSBBs) in a large cohort of patients with CSPH;(ii) identification of markers of hemodynamic response(iii) identification of factors potentially affecting the accuracy of PPG measurement.

DETAILED DESCRIPTION:
Specific Aim 1 To explore the correlation between endoscopic ultrasound (EUS)-guided portal pressure gradient (PPG) and hepatic venous pressure gradient (HVPG) in evaluation of hemodynamic response to non-selective beta blockers (NSBBs) in patients with advanced chronic liver disease and high risk varices. The investigators will perform EUS-PPG measurement and HVPG measurement at baseline and after NSBBs titration in enrolled patients. Hemodynamic response to medical therapy is defined as either a decrease in HVPG by >20% of the baseline value or an absolute value of HVPG < 12 mmHg after dose titration.

Correlation between PPG/HVPG values and development of portal hypertension-related gastrointestinal bleeding or liver- related events (ascites, spontaneous bacterial peritonitis, and hepatic encephalopathy) will be clinically assessed during follow-up with outpatients visits every 2-3 months.

Specific Aim 2 Identification of other markers of hemodynamic response to non selective beta blockers (NSBBs), with focus on elastography modifications and gut microbiota composition. To identify predictors of hemodynamic response, splenic and hepatic elastography measurement will performed at baseline and after NSBBs titration. In the same way the investigators will evaluate the gut microbiota before and after the start of therapy with NSBBs.

Specific Aim 3 Identification of factors potentially affecting the accuracy of PPG measurement. It is well-known that deep sedation may cause inaccurate HVPG values, while mild sedation with low dose midazolam does not modify the HVPG. In a subgroup of enrolled patients the investigators will perform PPG measurement with deep and mild sedation in order to investigate influence of deep sedation on PPG measurement accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed esophago-gastric varices or with high suspicion of CSPH at non-invasive tests (porto- systemic collaterals at imaging, platelet count <150.000 x mm3, spleen size >13 cm in the largest axis, alteration of elastography parameters of the liver or spleen)
* naïve to treatment with NSBBs,

Exclusion Criteria:

* Child Pugh >A6
* Hepatocellular carcinoma
* Portal vein thrombosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive outpatients with newly diagnosed esophago-gastric varices or with high suspicion of CSPH at non-invasive tests, naïve to treatment with NSBBs, will be evaluated over a two-years period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the portal pressure gradient though endoscopic ultrasound (EUS) and hepatic venous pressure gradient (HVPG) to evaluate the hemodynamic response to non-selective beta blockers (NSBBs) | 24 months
  The investigators will measure portal pressure gradient through EUS-PPG measurement at baseline and after NSBBs titration in enrolled patients.
HVPG Measurement Before and After NSBB Titration in Portal Hypertension | 24 months
  The investigators will measure portal pressure gradient through HVPG measurement at baseline and after NSBBs titration in enrolled patients.

SECONDARY OUTCOMES:
Markers of hemodynamic response | 24 months
  Spleen Stiffness Measurement (SSM) will be assessed by transient elastography before starting NSBB and using a FibroScan® (Echosens, Paris, France) after an overnight fasting.
Identifying Markers of Hemodynamic Response in Portal Hypertension | 24 months
  Liver Stiffness Measurement (LSM) will be assessed by transient elastography before starting NSBB and using a FibroScan® (Echosens, Paris, France) after an overnight fasting.
Clinical and Biochemical Indicators of Hemodynamic Response | 24 months
  The gut microbiota will be collected before and after the start of therapy with NSBBs. Fecal samples will be collected at home in a commercial sterile, dry screw-top container, and frozen at -80 °C within 24 hours, until further processing. Baseline and post NSBBs treatment blood samples collected from portal vein will be drawn, processed and stored at -80°C within 1 hour, until further processing.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Santopaolo, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS, Rome
Locations (1):
- Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided